CLINICAL TRIAL: NCT06775938
Title: Can Artificial Intelligence Take Place of Physical Medicine and Rehabilitation Physicians?: ChatGPT Versus Physical Medicine and Rehabilitation Residents
Brief Title: ChatGPT Versus Physical Medicine and Rehabilitation Residents
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Physiatrist, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 31.12.2024-2873
Record Dates: First submitted 2025-01-02; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Artificial Intelligence (AI); Resident Education
Keywords: Artificial Intelligence; ChatGPT; Educational Technology; Physical and Rehabilitation Medicine; Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Physical medicine and rehabilitation residents: The residents enrolled in the PMR specialization training program held throughout Turkey in May 2024
  Interventions: Other: resident exam
- ChatGPT: A new user was created for the free version of the ChatGPT-4o application, and a series of questions belonging to four distinct education levels were posed to it, one by one. For each question, ChatGPT was instructed to select only one option out of five.
  Interventions: Other: resident exam

INTERVENTIONS:
Other: resident exam — Resident exam in May 2024.

SUMMARY:
The aim of this study was to assess the performance of ChatGPT on examinations administered to physical medicine and rehabilitation (PMR) residents.

DETAILED DESCRIPTION:
These exams for resident physicians are annual exams administered throughout the training period, which constitute a fundamental component of the training process towards becoming a PMR physician. In this study, we evaluated the performance of ChatGPT in these exams, made separate assessments for each training year, and compared the results of ChatGPT with the results of residents who passed the same exam.

ELIGIBILITY:
Inclusion Criteria:

* Physical medicine and rehabilitation residents exam results in May 2024

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study used exam questions taken by the majority of residents enrolled in the PMR specialization training program held throughout Turkey in May 2024. These exam questions were selected from a pool of questions developed by lecturers affiliated with the PMR departments of hospitals affiliated with the University of Health Sciences. The exam questions were structured to cover four different difficulty levels.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
The comparison of resident exam results and ChatGPT answers to the same questions | through study completion, an average of 10 days
  In May 2024, the exam results of residents in training and research hospitals affiliated with the Health Sciences University across Türkiye will be compared with the answers and rankings given by ChatGPT to the same questions. ChatGPT accuracy rate and response time to questions will be determined. The minimum score to be obtained from this exam is 0 and the maximum score is 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided